CLINICAL TRIAL: NCT05971732
Title: The Effects of Ferric Derisomaltose Administered Before Hospital Discharge in Stabilised Patients With Acute Heart Failure and Iron Deficiency on Exercise Capacity and Quality of Life: a Randomised, Parallel-group, Double-blind, Placebo Controlled Trial (COREVIVE-HFrEF)
Brief Title: The Effects of Ferric Derisomaltose in Patients With Acute Heart Failure and Iron Deficiency on Exercise Capacity and Quality of Life(COREVIVE-HFrEF)
Acronym: COREVIVE-HFrEF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingyi Ren, Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Monofer-HFrEF
Record Dates: First submitted 2023-07-13; First posted 2023-08-02 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Iron Deficiency; Acute Heart Failure
Keywords: Exercise capacity; Quality of life; Acute Heart Failure
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric derisomaltose; Iron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric derisomaltose (Experimental): Iron to be administered as ferric derisomaltose.
  The treatment dose (mL) to be administered will be determined by the patient's body weight and hemoglobin (Hb) value.
  Where Hb ≥10 g/dL, dosage according to body weight is as follows:
  Body weight <50 kg: 20 mg/kg; Body weight 50 to <70 kg: 1000 mg; Body weight ≥70 kg: 20 mg/kg up to a maximum of 1500 mg.
  Where Hb <10 g/dL, dosage according to body weight is as follows:
  Body weight <50 kg: 20 mg/kg; Body weight 50 to <70 kg: 20 mg/kg; Body weight ≥70 kg: 20 mg/kg up to a maximum of 2000 mg.
  Infused over a minimum of 15mins for doses up to and including 1000mg, and a minimum of 30 mins for doses >1000mg
  Interventions: Drug: Ferric derisomaltose
- Placebo (Placebo Comparator): Participants in this arm will receive normal saline 0.9% in analogy to treatment arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric derisomaltose — After baseline assessments patients will be randomised in a 1:1 ratio to receive ferric derisomaltose IV or placebo (normal saline). In the Treatment group, Ferric derisomaltose will be administered according to the dosing schedule.
  Other Names: Monofer; Iron (III) isomaltoside 1000
  Arms: Ferric derisomaltose
Drug: Placebo — In the placebo group, patients will receive the equivalent number of normal saline injections.
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
This study will address whether the additional use of Ferric Derisomaltose on top of standard care will improve exercise capacity and quality of life in patients with acute heart failure and iron deficiency. One group of participants will receive treatment with Ferric Derisomaltose and the other group will receive normal saline 0.9% as placebo.

DETAILED DESCRIPTION:
Acute heart failure (AHF) is a very common medical problem. Despite improvements in treatment, many patients suffer limiting exercise capacity and quality of life. Previous comorbidities may account for it. Approximately 80% of patients hospitalized with AHF suffered from a combination of iron deficiency. A decline in exercise capacity may occur under this condition. Some research studies have suggested that giving CHF patients intravenous iron improves symptoms in the short term. It is unknown, however, whether correcting iron deficiency is beneficial to patients with AHF to improve excise capacity and whether it improves quality of life and accelerate recovery from acute duration. This study will help us answer these key questions.

This is an investigator-initiated, randomised, parallel group, double-blind, placebo-controlled trial, evaluating the excise capacity improvement of using ferric derisomaltose versus placebo in hospitalized patients with acute heart failure with reduced ejection fraction before discharge.

Participants will be assessed daily using 6-minute walking test after IV iron injection until discharge from hospital, especially focus on the change from baseline to the 3rd day. Some questionnaires are also conducted to evaluate the self-reported status. Participants will be followed up at 2 weeks and 4 weeks.

The primary and secondary endpoints will be examined in subgroups predefined by baseline variables reflecting demography, Hb level, etiology of HF, left ventricular ejection fraction, natriuretic peptide, index of iron metabolism, eGFR and others.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Clinical diagnosis of heart failure with reduced ejection fraction (HFrEF), defined as documented 2-dimensional echocardiography left ventricular ejection fraction (LVEF) <50% before randomization.
3. Currently hospitalised for an episode of acute heart failure (AHF) where AHF was the primary reason for hospitalisation, New York Heart Association (NYHA) class II - IV.
4. Reaching hemodynamic stability after standard treatment (if tolerated, initiate four pillars of guideline-directed medical therapies). All of the following (i.e., items a to c) must apply:

   1. Systolic blood pressure≥100mmHg, without symptoms of hypotension;
   2. Stop using intravenous diuretics;
   3. Neither intravenous inotropic drugs or vasodilators were used (including nitrates).
5. Subject is iron deficient defined as serum ferritin <100 ng/mL or 100 ng/mL ≤ serum ferritin ≤299 ng/mL if TSAT <20%.
6. Able and willing to provide informed consent and accomplish 6 minutes-walking test.

Exclusion Criteria:

1. Hematological criteria: ferritin >400 ug/L; hemoglobin <9.0, hemoglobin >13.5 g/dL in women or >14.5 g/dL in men.
2. Renal dialysis or MDRD/CKD-EPI estimated glomerular filtration rate (eGFR) <15ml/min/1.73m2
3. Body weight <35kg at randomization.
4. Heart failure was secondary to valvular diseases or congenital heart diseases.
5. History of acquired iron overload or hemochromatosis (or first-degree relative of hemochromatosis)
6. Known hypersensitivity reaction to any component of ferric derisomaltose (Monofer®) or any of its excipients (water for injections, sodium hydroxide (for pH adjustment), hydrochloric acid (for pH adjustment)).
7. Non-iron deficiency anaemia.
8. Already receiving erythropoiesis stimulating agents (ESA) or other iron supplements in previous 4 weeks prior to randomization.
9. Active infection (defined as currently treated with oral or intravenous antibiotics), bleeding (gastrointestinal haemorrhagia, menorrhagia, history of peptic ulcer with no evidence of healing or inflammatory bowel disease) and history of malignant tumor.
10. Any of the following diseases that hinders exercise testing: severe musculoskeletal disease, unstable angina, obstructive cardiomyopathy, severe uncorrected valvular disease, or uncontrolled slow or rapid arrhythmia (mean ventricular rate> 100 beats / min at rest).
11. Known positive HBsAg and/or HCV RNA; known HIV positivity; chronic liver disease (including active hepatitis), hepatic sclerosis, ALT or AST > 3x upper limit of normal.
12. Within 3 months of any of the following: acute myocardial infarction (AMI) or acute coronary syndrome (ACS), transient ischemic attack (TIA) or stroke, uncontrolled hypertension.
13. Revascularization therapy (coronary artery bypass grafting, percutaneous intervention, or major surgery) in the past 3 months; or planning cardiac surgery or revascularization.
14. Baseline 6 minutes-walking distance>500m.
15. Treated with long-term oral high-dose or steroid-immunosuppression therapy.
16. Investigator considers a possible alternative diagnosis to explain the patient's HF symptoms: severe obesity, primary pulmonary hypertension, or chronic obstructive pulmonary disease (COPD).
17. Subject is pregnant (e.g., positive human chorionic gonadotropin test) or breast feeding.
18. Untreated hypothyroidism.
19. Currently enrolled in any other investigational device or drug study <30 days prior to screening, or received other investigational agent(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walking distance | Up to 3 days
  The difference of 6-minute walking distance in meters from baseline to day3 after IV iron injection.

SECONDARY OUTCOMES:
Change From Baseline in 6-minute walking distance | At 2 weeks, 4weeks after IV iron injection
  The difference of 6-minute walking distance in meters from baseline at 2 weeks, 4weeks after IV iron injection.
Change From Baseline in the KCCQ Clinical Summary Score | At 2 weeks, 4weeks after IV iron injection
  KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ-clinical summary score was average of domains- physical limitation and total symptoms (average of symptom frequency and symptom burden), and transformed to a single score which ranged from 0 (worst) -100 (the best possible status), where the higher score reflected better health status.
Change From Baseline in the EQ-5D-5L Questionnaire Indexed Value | At 3 days, 2weeks, 4weeks after IV iron injection
  EQ-5D-5L: European Quality of Life-5 Dimensions-5 Levels The EQ 5D questionnaire consists of a health descriptive system for participants to self-classify and rate their health status on the day of administration.
  The descriptive system includes 5 items/dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, which are coded from 1 (best state) to 5 (worst state).
Change From Baseline in NYHA Functional Class | At 3 days, 2weeks, 4weeks after IV iron injection
  NYHA = New York Heart Association
  NYHA functional class was assessed as Class I, II, III, IV:
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest.
  Lower response categories are better for score NYHA.
Change From Baseline in PGA quality of life questionnaire | At 3 days, 2weeks, 4weeks after IV iron injection
  PGA:Patient Global Assessment
  PGA questionnaire consists of a health descriptive system for participants to self-reported and rate their medical condition after participate this study.
  The descriptive system includes 7 choices：has much improved, has (moderately) improved, has a little improved, is unchanged, is a little worse, is (moderately) worse, is much worse, which are coded from 1 (best state) to 7 (worst state).
Change From Baseline in Concentration of hemoglobin (Hb) | At 3 days, 2weeks, 4weeks after IV iron injection
  Hemoglobin (Hb) is a commonly used clinical test for assessing anaemia, with units of g/L.
Change From Baseline in proportion of reticulocyte (Ret%) | At 3 days, 2weeks, 4weeks after IV iron injection
  The reticulocyte ratio is often used to reflect the hematopoiesis of the bone marrow erythrocyte with units of percentage(%).
Change From Baseline in Concentration of ferritin | At 3 days, 2weeks, 4weeks after IV iron injection
  To assess the effect of ferric derisomaltose vs. placebo on change in ferritin from baseline to 3 days, 2weeks and 4weeks
Change From Baseline in concentration of transferrin saturation | At 3 days, 2weeks, 4weeks after IV iron injection
  To assess the effect of ferric derisomaltose vs. placebo on change in transferrin saturation from baseline to 3 days, 2weeks and 4weeks
Change From Baseline in Concentration of serum transferrin receptors (sTfR) | At 3 days, 2weeks, 4weeks after IV iron injection
  To assess the effect of ferric derisomaltose vs. placebo on change in serum transferrin receptors (sTfR) from baseline to 3 days, 2weeks and 4weeks
Change From Baseline in Concentration of N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) | At 3 days, 2weeks, 4weeks after IV iron injection
  To assess the effect of ferric derisomaltose vs. placebo on change in NT-proBNP from baseline to 3 days, 2weeks and 4weeks
Change From Baseline in Left Ventricular Systolic Function | At 2weeks, 4weeks after IV iron injection
  Left ventricular ejection fraction is assessed by two-dimensional directed M-mode echocardiography.
Change From Baseline in Left Ventricular End-Diastolic Diameter | At 2weeks, 4weeks after IV iron injection
  Left ventricular end-diastolic diameter is assessed by two-dimensional directed M-mode echocardiography.

OTHER OUTCOMES:
Change From Baseline in Urine Albumin-to-Creatinine Ratio (UACR) | At 3 days, 2weeks, 4weeks after IV iron injection
  Urine Albumin-to-Creatinine Ratio (UACR) is regard as a safety endpoint to reflect early injury of kidney.
A rise of high-sensitivity C-reaction protein (hs-CRP) levels from baseline | Up to 4weeks
  Safety endpoint is defined as a rise of high-sensitivity C-reaction protein (hs-CRP) from baseline.
Adverse Event after IV iron injection | Up to 4weeks
  Adverse Event Include Fishbane symptoms (flushing/chest pain/back pain/chest tightness, sometimes with dyspnea), isolated signs and symptoms (urticaria/pruritus/rash/mild hypotension, hypertension/tachycardia/nausea/headache), signs and symptoms of allergic reactions (persistent hypotension; airway angioedema/generalised urticaria, non-airway angioedema/wheezing, bronchospasm, vomiting, abdominal pain, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China